CLINICAL TRIAL: NCT03797131
Title: An Open Label Pilot Study to Evaluate the Effect of KB195, a Novel Prebiotic Gluco-Oligosaccharide Mixture, in the Diet of Patients With Urea Cycle Disorders on Gut Nitrogen Metabolism
Brief Title: Clinical Food Study to Evaluate the Effect of KB195 on Gut Nitrogen Metabolism in Patients With Urea Cycle Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K013-118
Record Dates: First submitted 2018-12-07; First posted 2019-01-09 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Urea Cycle Disorders
Keywords: KB195; Urea Cycle Disorders; UCD; microbiome; Kaleido; ammonia
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KB195 Arm (Experimental)
  Interventions: Other: KB195 (a novel mixture of oligosaccharides)

INTERVENTIONS:
Other: KB195 (a novel mixture of oligosaccharides) — KB195 (a novel mixture of oligosaccharides) for oral intake for 21 days.

SUMMARY:
This clinical food study aims to explore the effect of KB195, a novel mixture of oligosaccharides, on the metabolism of nitrogen by the microbiome in patients with urea cycle disorders (UCDs). This will be done using a stable isotope to assess nitrogen metabolism in the blood, urine, and stool. The study will also assess the safety and tolerability of KB195 in patients with UCDs.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed UCD patient at any age ≥ 14 years
* Parental/legal guardian permission or patient's written informed consent or assent, as applicable
* Be willing and able to comply with study requirements

Exclusion Criteria:

* Any medical condition unrelated to the sequelae of UCD
* Patient has N-acetylglutamate synthase (NAGS) deficiency
* Recent hospitalization or risk for metabolic decompensation
* Liver transplantation
* Systemic antibiotics, probiotics or prebiotics that do not align with study guidances
* Change in dose or frequency of any drug or other compound to modulate GI motility
* Contraindications or known allergy/sensitivity to the use of the study products
* Use of an investigational drug, product or device within 30 days prior to Screening Visit, or current enrolment in another investigational drug, product, or device study
* Considered to be at risk for noncompliance or unlikely for any reason to be able to comply with the study procedures

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in labelled (15N-nitrogen) and total nitrogen excretion in urine | Baseline to Day 25
  Evaluate the effect of KB195 on nitrogen metabolism in the gut of patients with UCD by analyzing the change in labelled (15N-nitrogen) and total nitrogen excretion in urine
Change in labelled (15N-urea) and total urea excretion in urine | Baseline to Day 25
  Evaluate the effect of KB195 on nitrogen metabolism in the gut of patients with UCD by analyzing the change in labelled (15N-urea) and total urea excretion in urine
Change in labelled (15N-ammonia) and total ammonia excretion in urine | Baseline to Day 25
  Evaluate the effect of KB195 on nitrogen metabolism in the gut of patients with UCD by analyzing the change in labelled (15N-ammonia) and total ammonia excretion in urine

SECONDARY OUTCOMES:
Change in Gastrointestinal Tolerability Questionnaire (GITQ) through the collection of daily patient questionnaires | Baseline to Day 32
  Evaluate the effect of KB195 on self-report questionnaires including the Gastrointestinal Tolerability Questionnaire, an assessment of the frequency and severity of GI symptoms, e.g., gas, abdominal pain, calculated on a scale from 0 (None/Not applicable) to a maximum score of 60 (Severe/Much more than usual) for all questions
Change in Bristol Stool Scale (BSS) through the collection of daily patient questionnaires | Baseline to Day 32
  Evaluate the effect of KB195 on self-report questionnaires including the Bristol Stool Scale, an assessment of stool consistency on a scale from 1 (separate hard lumps, like nuts, hard to pass) through 7 (watery, no solid pieces, entirely liquid).

OTHER OUTCOMES:
Incidence of adverse events | Baseline to Day 32

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, Study Director — Kaleido Biosciences
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No